CLINICAL TRIAL: NCT05980650
Title: The Effect of Reiki Administered to Risky Pregnant Women on Holistic Well-being, Prenatal, Maternal Attachment and Physical Symptoms: A Randomized Controlled Study
Brief Title: Reiki Effect on Risky Pregnants in Terms of Holistic Well-being, Prenatal, Maternal Attachment and Physical Symptoms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Dilara Keklik, Research Assistant, PhD, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 135
Record Dates: First submitted 2023-07-10; First posted 2023-08-08 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Pregnancy Complications
Keywords: reiki; Holistic Well-being; Maternal Attachment; Physical Symptoms
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reiki group (Experimental): Reiki will be implied to this group and this group will have routine nursing care given in the hospital during their hospitalization such as medical treatment implication and measuring vital signs
  Interventions: Other: Reiki implication
- Routine Nursing Care (No Intervention): This group will have just routine nursing care given in the hospital during their hospitalization such as medical treatment implication and measuring vital signs

INTERVENTIONS:
Other: Reiki implication — Reiki will be implicate by researcher by putting hands on patient
  Arms: Reiki group

SUMMARY:
Nurses should identify situations that may negatively affect mother-infant interaction from the prenatal period and mothers who experience these situations in order to ensure the establishment of secure attachment behavior. Then, they should cooperate with these mothers to eliminate negative situations or reduce their effects. It is also stated that practices such as meditation during pregnancy increase prenatal attachment.

Despite the benefits of Reiki application, no study has been found on the use of reiki in risky pregnant women. In this study, the effect of remotely applied reiki on high-risk pregnant women on holistic well-being, prenatal, maternal attachment and physical symptoms will be examined.

DETAILED DESCRIPTION:
Complications that occur in risky pregnancies that are not followed up and treated at regular intervals adversely affect maternal and fetal health, leading to outcomes that increase the risk of mortality and morbidity. As a matter of fact, it is seen that maternal deaths continue due to preventable or treatable causes during pregnancy or childbirth in the world and in our country. In addition, approximately 380 women become pregnant every minute in the world, half of them experience pregnancy-related complications and are classified in the risky pregnancy group.

The concept of well-being has emerged as a concept that further expands the views on health and gathers various health fields under one roof. Well-being is a subjective data reached by how individuals perceive their own lives. It is expressed in general judgments about affect and life satisfaction that change from joy to depression.

If pregnancy-related problems that negatively affect the perception of pregnancy are not managed well, it can cause psychological distress and reduce the level of psychological well-being of pregnant women. Psychological well-being is the positive psychological functioning of mental health. It is also expressed as the frequency of experiencing good or bad moods and emotions that have a positive or negative effect. Low level of psychological well-being during pregnancy is associated with many risks such as negative pregnancy outcomes, stress, anxiety, depression and behavioral problems in early childhood.

Attachment is defined as an instinctive process that serves to maintain closeness to the caregiver or as strong sensory bonds that people develop with people they deem important to them. In an other saying; Attachment is defined as the emotional bond between the child and his family. The tendency and need to establish emotional bonds are necessary for newborns to survive. Attachment can be prenatal and maternal attachment . He defined the mother's love for her baby during pregnancy and the bond she established with her as prenatal attachment. Prenatal attachment and adaptation to motherhood affect the baby's healthier growth and development and later on personality formation in childhood and adulthood. When there is a secure attachment during pregnancy, the woman realizes that her unborn baby has a relationship with her and sees her as a separate individual. This helps the expectant mother to show love and affection to her baby, to protect her, to feed her, to show interest, to interact and to be sensitive to her baby's needs, and facilitates the development of motherhood identity and adaptation to motherhood. A healthy maternal attachment process ensures a healthy communication between the mother and the baby, affects the baby's behavior positively, and gives happiness to the mother. As health professionals, nurses play an important role in the healthy development and maintenance of mother-infant attachment. If mother-infant bonding is not successful, the baby may experience physical, emotional, social, mental and language development problems. It is stated that the effects of secure or insecure attachment for mother and baby can last a lifetime. Attachment disorders can cause emotional disorders during pregnancy. In this respect, it is necessary to support expectant mothers with risky pregnancies where attachment may be affected.

The postpartum period is the harbinger of a new beginning for the woman and her family. During this period, important anatomical, physiological, psychological and endocrine changes are experienced in the mother's body. Depending on these changes, women experience a number of physical symptoms. In studies examining the physical symptoms experienced by women in the postpartum period; perineal problems, back pain, fatigue, pain in the incision/episiotomy area, headache, edema, hemorrhoids, constipation, urinary incontinence, sleep disturbance, sexual problems, painful coitus, and problems related to breastfeeding were determined to be common.

Reiki means "universal life energy". It is this universal, primary and creative source of power and energy that keeps us alive. Reiki is a natural healing energy. Reiki flows from the practitioner's hands in a powerful and concentrated way, making use of light and energy. It is a way of treating others physically and spiritually. Reiki focuses on energy chakras and bio-psycho-spiritual healing. Reiki allows vital signs (blood pressure, pulse rate, respiratory rate) to reach normal levels, reduces acute and chronic pain, facilitates sleep, reduces anxiety and fear, relieves depression, reduces stress, provides relaxation, reduces the use of painkillers, increases coping skills and facilitate communication.

ELIGIBILITY:
Inclusion Criteria:

* 28th and above gestational week,
* Having been diagnosed with a risky pregnancy,
* Able to read and write, • Open to communication,

Exclusion Criteria:

* Having a psychiatric history,
* Multiple pregnancy
* Giving a birth to a child with a chronic illness
* Women who have received energy therapies and reiki training such as Reiki touch therapy / Therapeutic touch / Healing touch before

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Risky pregnant women will be included in this study
Enrollment: 46 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Reiki effect on risky pregnants in terms of holistic well-being | postpartum 6th weeks
  Reiki may affect holistic well-being and holistic well-being scale points may be between 30 (minimum) and 300 (maximum) points in the postpartum 6th weeks. As the scale score approaches 300, holistic well-being increases and reaches a maximum at 300 points.
Reiki effect on risky pregnants in terms of prenatal attachment | change in prenatal attachment in 4 weeks
  Reiki may affect prenatal attachment and prenatal attachment scale points may be between 21 and 84 during prenatal period in 4 weeks. As the scale score approaches 84, prenatal attachment increases and reaches a maximum at 84. The increase in the score indicates that the attachment level of the pregnant also increases.
Reiki effect on risky pregnants in terms of postpartum physical symptoms | change in postpartum physical symptoms after giving a birth during 6 weeks
  Reiki may affect Postpartum Physical Symptom Severity which may be seen after giving a birth during 6 weeks. The minimum point is 0 and the maximum point is 54. It is expected to get score under 54 and close to 0 point from Postpartum Physical Symptom Severity Scale. The higher the score, the higher the postpartum physical symptom severity.
Reiki effect on risky pregnants in terms of maternal attachment | change in maternal attachment in the postpartum period in the sixth week
  Reiki may affect maternal attachment and maternal attachment scale points may become higher than 26 in the postpartum period in the sixth week. The highest score that can be obtained from the scale is 104, and the lowest score is 26. High scores mean good maternal attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Evşen Nazik, Study Director — Cukurova University
Locations (1):
- Adana City Hospital, Sariçam, Sa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be kept in confident